CLINICAL TRIAL: NCT04974112
Title: Multi-center Dynamic Investigation and Research on Nutritional Status of InpatientS
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Jinhua Central Hospital (Other); Huizhou Municipal Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-138
Record Dates: First submitted 2021-07-13; First posted 2021-07-23 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2015-05

CONDITIONS: Nutrition
Keywords: SGA NRS2002 nutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — 1. Newly hospitalized patients ≥ 18 years old;
  2. The length of hospital stay is 7-30 days;
  3. Those who have not undergone surgery before 8 o'clock the next day;
  4. Consciousness;
  5. Willing to accept the assessment and sign the informed consent form.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- General Surgery: This study was conducted in parallel in many Class-A hospitals across the country. Special researchers were assigned by the research unit to collect patient information using SGA and NRS2002 and other data measurement tools.
  Interventions: Other: Apply SGA and NRS2002
- Thoracic Surgery: This study was conducted in parallel in many Class-A hospitals across the country. Special researchers were assigned by the research unit to collect patient information using SGA and NRS2002 and other data measurement tools.
  Interventions: Other: Apply SGA and NRS2002
- orthopedics: This study was conducted in parallel in many Class-A hospitals across the country. Special researchers were assigned by the research unit to collect patient information using SGA and NRS2002 and other data measurement tools.
  Interventions: Other: Apply SGA and NRS2002
- Gastroenterology: This study was conducted in parallel in many Class-A hospitals across the country. Special researchers were assigned by the research unit to collect patient information using SGA and NRS2002 and other data measurement tools.
  Interventions: Other: Apply SGA and NRS2002
- Respiratory: This study was conducted in parallel in many Class-A hospitals across the country. Special researchers were assigned by the research unit to collect patient information using SGA and NRS2002 and other data measurement tools.
  Interventions: Other: Apply SGA and NRS2002
- Neurology: This study was conducted in parallel in many Class-A hospitals across the country. Special researchers were assigned by the research unit to collect patient information using SGA and NRS2002 and other data measurement tools.
  Interventions: Other: Apply SGA and NRS2002

INTERVENTIONS:
Other: Apply SGA and NRS2002 — Special researchers appointed by the research unit apply SGA and NRS2002 and other data measurement tools to collect patient information

SUMMARY:
we use the tools of SGA and NRS2002 to understand the nutritional status of Chinese Han inpatients during hospitalization and discharge, and to dynamically analyze the changes in the process of internal medicine and surgery in many general hospitals across Zhejiang Province.

DETAILED DESCRIPTION:
his study was conducted in parallel in a number of Grade-A hospitals across the country.

The researchers used SGA and NRS2002 and other data measurement tools to collect patient information.

1. General survey: initials, age, height, weight, gender, birthday, nationality;
2. Admission and discharge diagnosis: primary diagnosis and secondary diagnosis;
3. Laboratory indicators at admission and discharge: white blood cell, lymphocyte count, hemoglobin, platelet; Liver function (ALT and TBIL); kidney function (BUN and CR); protein (total protein, albumin and Prealbumin); blood lipids (cholesterol and triglycerides), etc.: The above results are subject to laboratory examinations within 3 days of hospitalization and discharge, and collect as complete as possible;
4. Anthropometric indicators at admission and discharge: hand grip, calf circumference or upper arm circumference, etc.
5. Comprehensive evaluation tools at admission and discharge: subjective comprehensive nutritional assessment (SGA) and nutritional risk screening (NRS2002);
6. Description of nutritional support during hospitalization: no nutritional support, pure enteral nutrition support, pure parenteral nutrition support, enteral + parenteral nutrition support;
7. Clinical outcome indicators at discharge: 30-day hospitalization mortality, total complications, infection complications, length of stay, total medical expenses, etc.

ELIGIBILITY:
Inclusion Criteria:

* Newly hospitalized patients ≥ 18 years old;
* The length of hospital stay is 7-30 days;
* Those who have not undergone surgery before 8 o'clock the next day;
* Consciousness;
* Willing to accept the assessment and sign the informed consent form.

Exclusion Criteria:

* Age <18 years old;
* The hospital stay is less than 7 days or more than 30 days;
* Those undergoing surgery before 8 o'clock the next day;
* Unconsciousness;
* Inpatients who refuse to be assessed.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatients in the hospital
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2014-04-20 (Actual); Primary Completion 2014-10-30 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
the nutritional status of Chinese Han inpatients during hospitalization and discharge | 2014-10
  Use NRS 2002 to understand the nutritional status of Chinese Han inpatients during hospitalization and discharge, and dynamically analyze the change process.

CONTACTS AND LOCATIONS:
Overall Officials: Fang He, MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hanzhong, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided